CLINICAL TRIAL: NCT03639168
Title: Chidamide Combined With Cisplatin in Recurrent or Metastatic Head and Neck Adenoid Cystic Carcinoma: A Prospective, Open-label, Phase II Study of a Single Center
Brief Title: Chidamide Combined With Cisplatin in Head and Neck Adenoid Cystic Carcinoma (HNACC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kai Xue, MD, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-HN-1
Record Dates: First submitted 2018-08-04; First posted 2018-08-21 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Adenoid Cystic Carcinomas; Cisplatin
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with Cisplatin (Experimental): Chidamide: 30mg,PO,biw one week before cycle 1 treatment Cisplatin 25mg/m2 ivgtt D1-3 Chidamide :20mg PO Biw, 2 week on , 1 week off
  Interventions: Drug: Chidamide combined with cisplatin

INTERVENTIONS:
Drug: Chidamide combined with cisplatin — Chidamide combined with cisplatin

SUMMARY:
The investigators conducted this study to evaluate the efficacy of Chidamide combined with cisplatin in recurrent or metastatic head and neck adenoid cystic carcinoma.

DETAILED DESCRIPTION:
Adenoid cystic carcinomas (ACCs) constitute of 1% of head and neck cancers. This type of tumor grows slowly with a high potential of local recurrence. Approximately 50% of patients develop distant metastases, and 33% patients die within 2 years. The initial therapy of these malignancies consists of surgical resection followed by radiotherapy. Systemic therapy is crucial in the management of recurrent and metastatic disease. However, nowadays, there were no standard chemoimmunotherapy regimes. Previous report showed that overall response rate was only less than 10% using single-agent chemotherapies, and the best results were achieved by cisplatin. Chidamide is a new benzamide class of histone deacetylase inhibitor with marked antitumor activity. And a phase I study has showed that one of three patients with submandibular adenoid cystic carcinoma achieved a partial response treated with Chidamide. The investigators conducted this study to evaluate the efficacy of Chidamide combined with cisplatin in recurrent or metastatic head and neck adenoid cystic carcinoma, in order to find a potential promising way to treat this kind of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75 years old
2. Histological confirmed recurrent or metastatic head and neck adenoid cystic carcinoma
3. Unable to treat with surgery/radiotherapy, or previously failure to non-cisplatin systematic treatment;
4. Eastern Cooperative Oncology Group performance status 0 to 2;
5. Patients have written informed consent to participate in the study;
6. anticipated to live ≧3 months;
7. Absolute neutrophil count ≥ 1.5×109/L，platelet ≥ 100×109/L，hemoglobin ≥ 90 g/L
8. total bilirubin < 1.5×upper limit of normal(ULN), ALT and AST < 3× ULN
9. serum creatine <1.5×ULN, and creatinine clearance rate (CCR) ≥ 50 ml/min
10. Ultrasonic cardiogram showed left ventricle ejection fraction ≥ 50%, EKG showed no signs of myocardial ischemia, with no previous arrhythmia which need pharmacological intervention.
11. Measurable disease was defined as at least one lesion ≥1.5 cm in length-diameter and ≥0.5 cm in short-diameter by CT.

Exclusion Criteria:

1. Previously treated with HDACi;
2. Treated with cisplatin-contained regimes in the past half of the year, and not achieving PR/CR;
3. History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix;
4. HIV, HCV, or syphilis infection；
5. Pregnant or lactating women;
6. Serious uncontrolled infection;
7. Severe neurol of mental illness, including dementia and epilepsy;
8. Having contraindications to the use of oral medication, such as unable to swallow, nausea and vomiting, chronic diarrhea or suffering from a bowel obstruction;
9. Participated in other clinical trials in 4 weeks;
10. Other coexisting diseases or situations that may cause patients to fail to complete clinical trials;
11. History of QTc interval prolongation (Male >450ms，Female >470ms), ventricular tachycardia, auricular fibrillation, heart block of more than II degrees, myocardial infarction in 1 year, congenital heart disease, with symptomatic coronary heart disease requiring medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 weeks
  Defined as numbers of patients achieved complete response and patial response of treatment

SECONDARY OUTCOMES:
Disease control rate (DCR) | 6 weeks
  Defined as numbers of patients achieved complete response, patial response, and stable disease of treatment
Progression-free survival (PFS) | 6 weeks
  Defined as the time from randomization until objective tumor progression or death
Scoring of quality of life: EORTC-QLQ-30 | 6 weeks
  Quality of life was evaluated using EORTC-QLQ-30. All subscales are summed to compute a total score, and total scores are recorded. Lower scores represent a better outcome.

OTHER OUTCOMES:
Serum ctDNA biomarker | throughout the treatment period，up to 6 months
  relationship between biomarker and treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kai Xue, MD, Principal Investigator — Department of medical oncology,Fudan University, Shanghai Cancer Center
Locations (1):
- Kai Xue, Shanghai, Shanghai Municipality, China